CLINICAL TRIAL: NCT01246531
Title: Clinical Investigation of Aging Men With Renal Stones: The Role of Bone Demineralization (Metabolic and Hormonal Assessment)
Brief Title: Metabolic Assessment of Aging Men With Urinary Lithiasis
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Eduardo Mazzucchi, University of São Paulo General Hospital
Other Study IDs: 0688/07
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-10

CONDITIONS: Urolithiasis and Aging; Renal Calcul and Metabolic Diseases; Urolithiasis and Osteoporosis
Keywords: Urolithiasis; Renal calculi; Aging; Osteoporosis
MeSH Terms: conditions — Urolithiasis; Metabolic Diseases; Osteoporosis; Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Urolithiasis: Case arm: men above fifty years-old with urolithiasis
- Control: Control arm: men above fifty years-old without urolithiasis

SUMMARY:
Urinary lithiasis is a common disease on young adults, but not so far on aging people. Nowadays, the investigators are seeing a gradative growth on men above sixty years old, mainly in industrialized countries. The purpose of this study is to investigate metabolic aspects of aging men with renal stones, towards blood tests, 24 hour-urinary samples, imagenological exams and bone densitometry. The investigators have made a case-control model.

DETAILED DESCRIPTION:
Urolithiasis is a common disease, with an overall prevalence about 2% in the world. Accordingly growth of life expectancy, elderly people become more susceptible to present renal calculi.

The investigators have two purposes: (1) evaluate metabolic disturbances in aging men with urinary lithiasis, and (2) evaluate bone demineralization in aging men with renal calculi.

The investigators have made a case-control model. The case-group is compposed by men with more than fifty years-old who had their first lithiasic diagnosis (renal colic ou incidental finding) after that age. The control-group is compposed by men with more than fifty years-old who had never diagnosed with renal stones. So the investigators have excluded men with repetitive episodes of renal colic, that could be negatively influence the outcomes of aging factors on urinary lithiasis. All the people have to submitted to blood tests, 24-hour urinary samples, abdominal ultrassonography and abdominal X-ray (or abdominal CT, if necessary); and bone densitometry. The investigators hope to achieve reliable conclusions about urinary lithogenesis.

Blood tests: total calcium, ionized calcium, uric acid, phosphorus, creatinine, urea, testosterone and parathyroid hormone.

24-hour urinary sample(s): calcium, uric acid, creatinine, citrate, sodium, pH and volume. Patients of the case arm had to collect 6 24-hour urine samples, while the control arm had collected 3 24-hour urine samples.

Data were analyzed using the Fischer's exact, Chi-square and Mann-Whitney tests; a level of significance of 5% was adopted.

ELIGIBILITY:
Inclusion Criteria:

* Men above fifty years-old with urolithiasis diagnosis (case arm)
* Men above fifty years-old without urolithiasis diagnosis (control arm)

Exclusion Criteria:

* Urolithiasis diagnosis (clinical or incidental) before fifty years-old.
* Urinary culture positive

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from Urological Division of University of São Paulo General Hospital, in São Paulo (Brazil). Towards data bank, we called patients above fifty years-old who had urolithiasis diagnosis. Patients with benign prostate hyperplasia, above fifty years-old, had called to the control group.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Hypocitraturia is the main metabolic disturbance in aging men with urinary lithiasis | Two years
  Aging men that had initiated their clinical signs or symptoms of urinary lithiasis above fifty years-old, presented hypocitraturia like the most common metabolic disturbance in 24-hour urine analysis. This finding had been different when we look for younger renal stones formers. In these, hypercalciuria is the main metabolic disturbance. Idiopathic hypercalciuria could affect men in a precocious phase of their lives, because of the genetic basis. However hypocitraturia could be related with acidified status, secondarily to alimentary habits, mainly excessive protein and sodium diarily intake.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Mazzucchi, MD, Principal Investigator — University of São Paulo General Hospital - Division of Urology
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Usui Y, Matsuzaki S, Matsushita K, Shima M. Urolithiasis in geriatric patients. Tokai J Exp Clin Med. 2003 Jul;28(2):81-7. PMID 14714833
- [Background] Vella M, Karydi M, Coraci G, Oriti R, Melloni D. Pathophysiology and clinical aspects of urinary lithiasis. Urol Int. 2007;79 Suppl 1:26-31. doi: 10.1159/000104438. PMID 17726349
- [Background] Ebeling PR. Clinical practice. Osteoporosis in men. N Engl J Med. 2008 Apr 3;358(14):1474-82. doi: 10.1056/NEJMcp0707217. No abstract available. PMID 18385499
- [Background] Aw D, Silva AB, Palmer DB. Immunosenescence: emerging challenges for an ageing population. Immunology. 2007 Apr;120(4):435-46. doi: 10.1111/j.1365-2567.2007.02555.x. Epub 2007 Feb 15. PMID 17313487
- [Derived] Freitas Junior CH, Mazzucchi E, Danilovic A, Brito AH, Srougi M. Metabolic assessment of elderly men with urolithiasis. Clinics (Sao Paulo). 2012;67(5):457-61. doi: 10.6061/clinics/2012(05)09. PMID 22666789